CLINICAL TRIAL: NCT02513485
Title: "Inflammation-related Alterations in Neurocircuitry: Reversal With Levodopa"; "Inflammation Effects on Corticostriatal Connectivity and Reward: Role of Dopamine"
Brief Title: Inflammation-related Alterations in Neurocircuitry: Reversal With Levodopa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jennifer Felger, Associate Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00081486; R01MH109637 (NIH)
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Results first posted 2022-05-17 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-08

CONDITIONS: Depression
Keywords: Inflammation; Anhedonia; Psychomotor retardation
MeSH Terms: conditions — Depression; Inflammation; Anhedonia; Psychomotor Disorders | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sinemet/Placebo (Active Comparator): Subjects with major depression will be given Sinemet (a combination of 250 mg of levodopa and 50 mg of carbidopa) at one study visit and placebo at the other study visit. Sinemet will be given first followed by placebo at the subsequent visit.
  Interventions: Drug: Levodopa+carbidopa; Drug: Placebo
- Placebo/Sinemet (Active Comparator): Subjects with major depression will be given placebo at one study visit and Sinemet (a combination of 250 mg of levodopa and 50 mg of carbidopa) at the other study visit. Placebo will be given first followed by Sinemet at the subsequent visit.
  Interventions: Drug: Levodopa+carbidopa; Drug: Placebo

INTERVENTIONS:
Drug: Levodopa+carbidopa — Sinemet is a combination of 250 mg levodopa and 50 mg carbidopa. Sinemet will be administered orally at Visit 1 or Visit 2.
  Other Names: Sinemet
Drug: Placebo — A placebo is a sugar pill that has no therapeutic effect and will be administered orally at Visit 1 or Visit 2.

SUMMARY:
The purpose of this study is to learn more about the changes that happen in the brain and the body when a person is depressed. This study will determine if the level of inflammation in the body is related to symptoms of depression, how well the person thinks, and how certain brain regions communicate.

DETAILED DESCRIPTION:
Cytokines released by an activated immune system have been associated with decreased brain dopamine and the development of depression. Biomarkers of inflammation, such as inflammatory cytokines and acute-phase proteins like C-reactive protein (CRP), are elevated in a significant proportion of patients with mood and psychiatric disorders. The investigators will study if administration of Levodopa (L- 3,4-dihydroxyphenylalanine [DOPA]-carbidopa, 250/25mg) to depressed patients with high inflammation will 1) increase corticostriatal functional connectivity, and 2) improve objective measures of motivation compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have signed a current version of the Informed Consent and HIPAA documents prior to initiation of study procedures
* Able to comprehend English
* Diagnosis of Diagnostic and Statistical Manual of Mental Disorders (DSM)-V major depression and currently off antidepressant medication, unless otherwise approved by the PI or PI's designee
* Depression as the primary axis I disorder
* Negative pregnancy test for women of childbearing potential
* Not breast feeding
* At least two CRP tests conducted to establish reliability

Exclusion Criteria:

* Evidence of untreated or poorly controlled endocrine, cardiovascular, pulmonary, hematological, renal, or neurological disease
* History of central nervous system (CNS) trauma or active seizure disorder requiring medication unless otherwise approved by principal investigator, or PI's designee
* Current or history of migraines, glaucoma, melanoma, or bleeding disorder of any kind
* Autoimmune or inflammatory disorder of any kind
* Embedded metallic objects, prosthetics made of paramagnetic metals, aneurysmal clips and/or a history of claustrophobia
* Chronic infection (e.g. hepatitis B or C or Human Immunodeficiency Virus infection)
* Chronic use of agents known to affect the immune system including glucocorticoid therapy within the past 6 months, methotrexate within the past 1 year, chemotherapy of any kind (past or present), immunotherapy of any kind (past or present), aspirin or non-steroidal anti-inflammatory drugs (NSAIDs; within the past 2 weeks), statins (within the past 1 month), vaccinations (within the past 2 weeks), topical steroids (within the past 2 weeks), and antibiotics (within the past two weeks) unless otherwise approved by principal investigator or PI's designee.
* Suicide attempt within six months of screening, or active suicidal intent or plan, or score >2 on Hamilton Depression Rating Scale (HDRS), or Quick Inventory of Depressive Symptomatology Self-Report (QIDS) or Patient Health Questionnaire (PHQ-9) Suicide Item, unless otherwise approved by the PI or PI's designee
* A positive pregnancy test
* Organ transplants
* Current or history of cancer within the past five years besides basal cell carcinoma, unless otherwise approved by the PI or PI's designee
* A score of <28 on the Mini Mental Status Exam (MMSE), unless otherwise approved by the PI or PI's designee
* Wide Range Achievement Test (WRAT-3) score indicating less than 8th grade reading level, unless otherwise approved by the PI or PI's designee
* Either QIDS <14 or PHQ-9 <15, or HDRS <18, unless otherwise approved by the principal investigator or PI's designee
* History of the following: schizophrenia, schizoaffective disorder, other (non mood disorder) psychosis, depression secondary to a medical condition, mental retardation, dementia, or delirium
* Substance dependence [or abuse within the past year (except nicotine)], unless otherwise approved by the PI or PI's designee
* Body Mass Index >40 to limit the impact of morbid obesity on the results, unless otherwise approved by the principal investigator or PI's designee
* Antisocial personality disorder diagnosis as assessed during clinical interview, as well as a history of hospitalization and/or recurrent suicidal behavior judged to be directly due to the personality disorder
* Current eating disorder (except binge eating related to depression) unless approved by PI or PI's designee
* Current obsessive-compulsive disorder (OCD), exclusionary only if impacting daily functioning, as assessed by clinical interview
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with participating in or completing the protocol
* Smoking more than 1/2 pack a day or e-cigarette equivalent, unless approved by the PI or PI's designee
* Initiation of any of the following medications, unless otherwise approved by the PI or PI's designee: Aspirin or Aspirin-like compounds, Ibuprofen or Naproxen Sodium, Cholesterol medications, Antibiotics, Herbal Medications, Psychiatric or Psychotropic Medications, Omega-3 supplements, Topical Steroids, Vaccinations
* Currently on antidepressant medication, unless otherwise approved by the PI or PI's designee

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-10-09 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Felger, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bekhbat M, Li Z, Mehta ND, Treadway MT, Lucido MJ, Woolwine BJ, Haroon E, Miller AH, Felger JC. Functional connectivity in reward circuitry and symptoms of anhedonia as therapeutic targets in depression with high inflammation: evidence from a dopamine challenge study. Mol Psychiatry. 2022 Oct;27(10):4113-4121. doi: 10.1038/s41380-022-01715-3. Epub 2022 Aug 4. PMID 35927580

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between October 2015 and February 2020.
Groups:
- Sinemet/Placebo: Subjects with major depression were given Sinemet (a combination of 250 mg of levodopa and 50 mg of carbidopa) at one study visit and placebo at the other study visit. Sinemet was given first followed by placebo at the subsequent visit.
  Levodopa+carbidopa: Sinemet is a combination of 250 mg levodopa and 50 mg carbidopa. Sinemet was administered orally at Visit 1 or Visit 2.
  Placebo: A placebo is a sugar pill that has no therapeutic effect and was administered orally at Visit 1 or Visit 2.
- Placebo/Sinemet: Subjects with major depression were given placebo at one study visit and Sinemet (a combination of 250 mg of levodopa and 50 mg of carbidopa) at the other study visit. Placebo was given first followed by Sinemet at the subsequent visit.
  Levodopa+carbidopa: Sinemet is a combination of 250 mg levodopa and 50 mg carbidopa. Sinemet was administered orally at Visit 1 or Visit 2.
  Placebo: A placebo is a sugar pill that has no therapeutic effect and was administered orally at Visit 1 or Visit 2.
Period: Overall Study
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Started | 28 | 29
Completed | 27 | 29
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sinemet/Placebo | Placebo/Sinemet | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (11.5) | 38.7 (10.3) | 37.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 26 | 24 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 8 | 23
  White | 11 | 20 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Corticostriatal Connectivity
Description: Corticostriatal connectivity was assessed by functional magnetic resonance imaging (fMRI). Resting-state and task-based (monetary incentive delay [MID]) fMRI scans were conducted on a 3 Tesla Siemens Trio MRI scanner. Subject-level correlations for degree of cortical and striatal functional connectivity were Fisher's Z transformed {Z(R)=0.5ln[(1+R)/(1-R)]}, a standard method for calculating fMRI functional connectivity. Greater Fisher's Z-scores reflected stronger correlated fMRI activity (i.e., higher corticostriatal connectivity).
Time Frame: Scans approximately 45 min post drug/placebo administration at Visit 1, Visit 2 (spaced by approximately 1 week)
Population: The number analyzed in one or more rows correspond to the number with available and analyzable resting fMRI scans both pre and post drug and placebo.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 21 | 19
Z-score
  Visit 1 resting corticostriatal connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  Visit 1 resting corticostriatal connectivity response to drug/placebo (post minus pre) | 0.10 (0.22) | 0.04 (0.17)
  Visit 2 resting corticostriatal connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  Visit 2 resting corticostriatal connectivity response to drug/placebo (post minus pre) | 0.07 (0.18) | 0.00 (0.23)
  Visit 1 resting corticostriatal connectivity post drug/placebo | 0.22 (0.15) | 0.24 (0.12)
  Visit 2 resting corticostriatal connectivity post drug/placebo | 0.24 (0.18) | 0.17 (0.18)
  Visit 1 task (reward anticipation) corticostriatal connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  Visit 1 task (reward anticipation) corticostriatal connectivity post drug/placebo | 0.02 (0.16) | 0.00 (0.15)
  Visit 2 task (reward anticipation) corticostriatal connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  Visit 2 task (reward anticipation) corticostriatal connectivity post drug/placebo | -0.04 (0.19) | -0.03 (0.16)

2. Primary Outcome: Correlation Coefficient Between Change in Corticostriatal Connectivity and Levels of Plasma C-reactive Protein and Other Immune Markers
Description: Peripheral blood samples were analyzed for levels of immune markers like plasma C-reactive protein (CRP), interleukin-6 (IL-6), soluble interleukin-6 receptor (sIL-6R), tumor necrosis factor (TNF) -alpha, soluble cytokine receptor2 (TNFR 2), interleukin-1 beta (IL-1 beta), interleukin-1 receptor antagonist (IL-1Ra), interleukin 10 (IL-10) and monocyte chemoattractant protein-1 (MCP-1).
Time Frame: Scans approximately 45 minutes post drug/placebo administration at Visit 1, Visit 2 (spaced by approximately 1 week)
Population: The number analyzed in each row correspond to the number available and analyzable with resting fMRI scans both pre and post drug and placebo.
Measure: Number (95% Confidence Interval); unit: Pearson's r Correlation Coefficient
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 21 | 19
Pearson's r Correlation Coefficient
  CRP mg/L and Visit 1 resting connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  CRP mg/L and Visit 1 resting connectivity response to drug/placebo (post minus pre) | 0.36 [-0.16 to 0.73] | -0.15 [-0.61 to 0.40]
  CRP mg/L and Visit 2 resting connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  CRP mg/L and Visit 2 resting connectivity response to drug/placebo (post minus pre) | -0.12 [-0.58 to 0.40] | 0.44 [-0.09 to 0.78]
  CRP mg/L and Visit 1 resting connectivity post drug/placebo | 0.10 [-0.35 to 0.51] | 0.15 [-0.33 to 0.56]
  CRP mg/L and Visit 2 resting connectivity post drug/placebo | -0.10 [-0.51 to 0.35] | 0.41 [-0.06 to 0.73]
  CRP mg/L and Visit 1 task (reward anticipation) connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  CRP mg/L and Visit 1 task (reward anticipation) connectivity post drug/placebo | 0.49 [-0.01 to 0.79] | -0.31 [-0.71 to 0.25]
  CRP mg/L and Visit 2 task (reward anticipation) connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  CRP mg/L and Visit 2 task (reward anticipation) connectivity post drug/placebo | 0.10 [-0.42 to 0.57] | 0.25 [-0.30 to 0.68]
  CRP > vs. < 2 mg/ and Visit 1 resting connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  CRP > vs. < 2 mg/ and Visit 1 resting connectivity response to drug/placebo (post minus pre) | 0.20 [-0.32 to 0.64] | 0.04 [-0.48 to 0.54]
  CRP > vs. < 2 mg/L and Visit 2 resting connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  CRP > vs. < 2 mg/L and Visit 2 resting connectivity response to drug/placebo (post minus pre) | -0.33 [-0.71 to 0.20] | 0.52 [0.01 to 0.81]
  CRP > vs. < 2 mg/L and Visit 1 resting connectivity post drug/placebo | 0.12 [-0.33 to 0.53] | 0.17 [-0.31 to 0.58]
  CRP > vs. < 2 mg/L and Visit 2 resting connectivity post drug/placebo | -0.31 [-0.66 to 0.14] | 0.38 [-0.09 to 0.71]
  CRP > vs. < 2 mg/L and Visit 1 task (reward anticipation) connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  CRP > vs. < 2 mg/L and Visit 1 task (reward anticipation) connectivity post drug/placebo | 0.22 [-0.31 to 0.65] | -0.35 [-0.73 to 0.20]
  CRP > vs. < 2 mg/L and Visit 2 task (reward anticipation) connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  CRP > vs. < 2 mg/L and Visit 2 task (reward anticipation) connectivity post drug/placebo | -0.18 [-0.62 to 0.35] | 0.48 [-0.05 to 0.80]
  Sum of cytokine Z scores and Visit 1 resting connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  Sum of cytokine Z scores and Visit 1 resting connectivity response to drug/placebo (post minus pre) | 0.40 [-0.12 to 0.75] | -0.05 [-0.56 to 0.49]
  Sum of cytokine Z scores and Visit 2 resting connectivity response to drug/placebo (post minus pre): number analyzed (Participants) | 16 | 15
  Sum of cytokine Z scores and Visit 2 resting connectivity response to drug/placebo (post minus pre) | -0.14 [-0.58 to 0.39] | 0.29 [-0.29 to 0.71]
  Sum of cytokine Z scores and Visit 1 resting connectivity post drug/placebo | 0.15 [-0.30 to 0.55] | -0.05 [-0.57 to 0.49]
  Sum of cytokine Z scores and Visit 2 resting connectivity post drug/placebo | -0.22 [-0.60 to 0.23] | 0.08 [-0.40 to 0.53]
  Sum of cytokine Z scores and Visit 1 task (reward anticipation) connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  Sum of cytokine Z scores and Visit 1 task (reward anticipation) connectivity post drug/placebo | 0.26 [-0.27 to 0.67] | -0.34 [-0.74 to 0.23]
  Sum of cytokine Z scores and Visit 2 task (reward anticipation) connectivity post drug/placebo: number analyzed (Participants) | 16 | 15
  Sum of cytokine Z scores and Visit 2 task (reward anticipation) connectivity post drug/placebo | 0.04 [-0.45 to 0.53] | -0.18 [-0.65 to 0.39]

3. Secondary Outcome: Effort-Expenditure for Rewards Task (EEfRT) Neurocognitive Test
Description: The Effort-Expenditure for Rewards Task (EEfRT) is a computer-based multi-trial task used to objectively assess motivation. Possible results range between 0 to1 with 1 being a better outcome. Results show mean probability of hard (high effort) choice.
Time Frame: At baseline and approximately 2-3 hours post drug/placebo administration at Visit 1, Visit 2 (spaced by approximately 1 week)
Population: This analysis includes participants who completed this assessment and had usable data. Two participants in each study arm did not complete this assessment at any time point. Two participants in the Placebo/Sinemet group had unusable data for the baseline assessment.
Measure: Mean (Standard Deviation); unit: Probability of hard/high effort choices
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 25 | 27
Probability of hard/high effort choices
  Baseline Visit (Task Practice): number analyzed (Participants) | 25 | 25
  Baseline Visit (Task Practice) | 0.29 (0.13) | 0.39 (0.17)
  Visit 1: 2-3 hrs post drug/placebo | 0.28 (0.13) | 0.34 (0.17)
  Visit 2: 2-3 hrs post drug/placebo | 0.30 (0.15) | 0.34 (0.21)

4. Secondary Outcome: The Trail Making Test (TMT) Neurocognitive Assessment
Description: The Trail Making Test (TMT) is used to measure basic attention and psychomotor processing speed. Time taken to complete each task is recorded in seconds, whereby the greater the number of seconds, the slower the psychomotor speed.
Time Frame: as for outcome 3
Population: This analysis includes participants who completed this assessment and had usable data. One participant in the Sinemet/Placebo arm and two participants in the Placebo/Sinemet arm did not complete this assessment at any time point. Three participants in the Placebo/Sinemet group had unusable data for the baseline assessment.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 26 | 27
seconds
  Baseline Visit (Task Practice): number analyzed (Participants) | 26 | 24
  Baseline Visit (Task Practice) | 24.0 (10.0) | 23.7 (4.7)
  Visit 1: 2-3 hrs post drug/placebo | 21.7 (8.8) | 21.0 (5.2)
  Visit 2: 2-3 hrs post drug/placebo | 23.0 (13.8) | 19.7 (4.6)

5. Secondary Outcome: Digit Symbol Task Neurocognitive Test
Description: The Digit Symbol Task was used to assess graphomotor speed, visual scanning and memory processing speed involving numbers and a corresponding blank box where subjects are asked to fill in matching symbol as fast as they can. Results show the average number of correct symbols completed in up to 100 boxes in 90 seconds.
Time Frame: as for outcome 3
Population: This analysis includes participants who completed this assessment and had usable data. One participant in the Placebo/Sinemet arm did not complete this assessment at any time point and one had unusable data for the baseline assessment.
Measure: Mean (Standard Deviation); unit: number of correct symbols
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 27 | 28
number of correct symbols
  Baseline Visit (Task Practice): number analyzed (Participants) | 27 | 27
  Baseline Visit (Task Practice) | 52.0 (8.8) | 54.9 (11.3)
  Visit 1: 2-3 hrs post drug/placebo | 61.3 (11.3) | 64.5 (10.2)
  Visit 2: 2-3 hrs post drug/placebo | 66.6 (11.7) | 66.4 (11.6)

6. Secondary Outcome: Finger Tapping Task (FTT) Neurocognitive Test
Description: The Finger Tapping Task (FTT) assesses motor speed and can detect subtle motor impairment. The test measures the average number of taps per 10 second trial. A greater number of taps reflects faster motor speed.
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of taps
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 27 | 28
number of taps
  Baseline Visit (Task Practice): number analyzed (Participants) | 27 | 27
  Baseline Visit (Task Practice) | 52.0 (8.8) | 54.9 (11.3)
  Visit 1: 2-3 hrs post drug/placebo | 61.3 (11.3) | 64.5 (10.2)
  Visit 2: 2-3 hrs post drug/placebo | 66.6 (11.7) | 66.4 (11.6)

7. Secondary Outcome: Reaction Time Task (CANTAB) Neurocognitive Test
Description: The reaction time test includes simple and choice reaction time tasks and is divided into 5 stages requiring increasingly complex chains of responses. The task provided distinction between reaction (or decision) time and movement latencies (milliseconds) based on touch responses made to a single (simple) or chosen from multiple (choice) stimuli flashed on a computer screen. Results show mean response latency in milliseconds.
Time Frame: as for outcome 3
Population: This analysis includes participants who completed this assessment and had usable data. Seven participants in the Sinemet/Placebo arm and 8 participants in the Placebo/Sinemet arm did not complete this assessment at any time point. One participant in each study arm had unusable data for the baseline assessment.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 20 | 21
milliseconds
  Baseline Simple Motor Time: number analyzed (Participants) | 19 | 20
  Baseline Simple Motor Time | 266.92 (59.55) | 276.12 (94.35)
  Baseline Choice Motor Time: number analyzed (Participants) | 19 | 20
  Baseline Choice Motor Time | 286.82 (50.47) | 299.57 (89.33)
  Baseline Simple Reaction Time: number analyzed (Participants) | 19 | 20
  Baseline Simple Reaction Time | 360.84 (38.38) | 356.53 (42.11)
  Baseline Choice Reaction Time: number analyzed (Participants) | 19 | 20
  Baseline Choice Reaction Time | 397.60 (46.74) | 394.82 (31.31)
  Visit 1: 2-3 hrs post drug/placebo Simple Motor Time | 240.62 (55.50) | 258.53 (89.29)
  Visit 1: 2-3 hrs post drug/placebo Choice Motor Time | 268.69 (52.17) | 284.94 (75.16)
  Visit 1: 2-3 hrs post drug/placebo Simple Reaction Time | 256.99 (35.69) | 348.93 (26.14)
  Visit 1: 2-3 hrs post drug/placebo Choice Reaction Time | 397.07 (39.50) | 385.03 (22.59)
  Visit 2: 2-3 hrs post drug/placebo Simple Motor Time | 241.28 (46.34) | 268.37 (93.51)
  Visit 2: 2-3 hrs post drug/placebo Choice Motor Time | 260.47 (42.43) | 296.94 (83.62)
  Visit 2: 2-3 hrs post drug/placebo Simple Reaction Time | 358.59 (35.87) | 361.76 (47.55)
  Visit 2: 2-3 hrs post drug/placebo Choice Reaction Time | 395.22 (33.75) | 396.68 (38.93)

8. Secondary Outcome: Multidimensional Fatigue Inventory (MFI) Self-report Questionnaire
Description: The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure severity of fatigue based on five dimensions of fatigue, general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. The total MFI scores range from 20 to 100 where high scores indicate greater fatigue.
Time Frame: At baseline and Visit 1, Visit 2 (spaced by approximately 1 week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 27 | 29
score on a scale
  Baseline | 74.7 (10.9) | 72.7 (13.5)
  Visit 1: Pre drug/placebo | 76.7 (10.7) | 74.2 (15.05)
  Visit 2: Pre drug/placebo | 75.7 (10.5) | 74.1 (14.9)

9. Secondary Outcome: Snaith-Hamilton Pleasure Scale (SHAPS) Self-report Questionnaire
Description: The Snaith-Hamilton Pleasure Scale (SHAPS), a 14-item self-report scale with high psychometric validity for assessing the presence of anhedonia, was used to assess hedonic capacity. Participants rated how much they agreed or disagreed with the 14 items phrased as "I would enjoy __" based on their ability to experience pleasure. Of the four possible response categories (Definitely Agree, Agree, Disagree, and Strongly Disagree), either of the Disagree responses received a score of 1 and either of the Agree responses received a score of 0. The SHAPS score calculated as the sum of these 14 items ranged from 0 to 14, and higher SHAPS scores indicated greater anhedonia.
Time Frame: Visit 1: Pre drug/placebo, Visit 1: 1-2 hrs post drug/placebo, Visit 2: Pre drug/placebo, Visit 2: 1-2 hrs post drug/placebo
Population: This analysis includes participants who completed this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 27 | 28
score on a scale
  Visit 1: Pre drug/placebo | 4.7 (3.5) | 5.8 (3.7)
  Visit 1: 1-2 hrs post drug/placebo | 4.3 (4.0) | 4.6 (3.7)
  Visit 2: Pre drug/placebo | 4.2 (3.9) | 4.9 (4.2)
  Visit 2: 1-2 hrs post drug/placebo | 4.2 (4.4) | 3.9 (4.2)

10. Secondary Outcome: Inventory of Depressive Symptoms-Self Report (IDS-SR) Questionnaire
Description: The Inventory of Depressive Symptoms-Self Report (IDS-SR) is a 30-item self-report instrument with excellent psychometric properties for measuring symptom constructs consistent with current Diagnostic and Statistical Manual of Mental Disorders (DSM) nosology and that is widely used to measure depression severity in clinical trials. Response scores are summed and range from 0 to 84, with higher scores reflecting greater depression severity.
Time Frame: At baseline and Visit 1: Pre drug/placebo, Visit 2: Pre drug/placebo (spaced by approximately 1 week)
Population: Three participants in the Sinemet/Placebo arm and four participants in the Placebo/Sinemet arm had unusable data for the baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 27 | 29
score on a scale
  Baseline: number analyzed (Participants) | 24 | 25
  Baseline | 37.9 (65) | 35.0 (10.8)
  Visit 1: Pre drug/placebo | 37.6 (6.3) | 31.8 (10.7)
  Visit 2: Pre drug/placebo | 34.7 (8.6) | 32.0 (11.1)

11. Secondary Outcome: Beck Depression Inventory (BDI-II), Anhedonia Subscale Score
Description: The Beck Depression Inventory-II (BDI-II) is a widely used self-report for measuring depression severity over the past two weeks and the anhedonia subscale is one of several validated subscales in the BDI-II. Responses are given on a 4-point scale where 0 = the symptom of depression has not been experienced and 3 = the symptom of depression is severe. The anhedonia subscale score is created by summing responses to four items of the BDI-II that assess loss of pleasure, loss of interest, loss of energy, loss of sex drive. The total score of the anhedonia subscale ranges from 0 to 12 where higher scores reflect greater severity of anhedonia symptoms.
Time Frame: Visit 1: Pre drug/placebo, Visit 2: Pre drug/placebo (spaced by approximately 1 week)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 27 | 29
score on a scale
  Visit 1: Pre drug/placebo | 6.4 (2.4) | 5.9 (2.5)
  Visit 2: Pre drug/placebo | 5.7 (2.9) | 5.9 (2.8)

12. Secondary Outcome: Profile of Mood States (POMS) Scale
Description: The Profile of Mood States (POMS) scale is a 30-item psychological rating scale used to assess transient, distinct mood states. Participants rate the extent to which they feel unhappy, blue, lonely, gloomy, and worthless on a scale from 0 (not at all) to 4 (extremely). Scores range from 0 to 120 with higher scores reflecting a more negative mood state.
Time Frame: as for outcome 9
Population: This analysis includes participants who completed this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 25 | 26
score on a scale
  Visit 1: Pre drug/placebo | 60.2 (17.6) | 57.0 (14.6)
  Visit 1: 1-2 hrs post drug/placebo | 54.0 (15.1) | 51.5 (11.8)
  Visit 2: Pre drug/placebo | 53.0 (12.7) | 56.2 (14.3)
  Visit 2: 1-2 hrs post drug/placebo | 48.5 (14.3) | 51.0 (11.5)

13. Secondary Outcome: State-Trait Anxiety Inventory (STAI) State Scale
Description: The 20-item self-report State-Trait Anxiety Inventory (STAI) State scale was used to measure severity of anxiety symptoms. Total scores range from 20 to 80 with higher scores reflecting greater anxiety. Scores in the high 40s are considered clinically significant.
Time Frame: as for outcome 9
Population: This analysis includes participants who completed this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 14 | 16
score on a scale
  Visit 1: Pre drug/placebo | 52.1 (12.3) | 46.5 (10.6)
  Visit 1: 1-2 hrs post drug/placebo | 49.2 (9.3) | 42.2 (9.3)
  Visit 2: Pre drug/placebo | 51.3 (9.9) | 45.9 (14.0)
  Visit 2: 1-2 hrs post drug/placebo | 43.4 (12.0) | 43.0 (9.9)

14. Secondary Outcome: Change in Motivation and Pleasure (MAP) Scale Score
Description: The motivation and pleasure (MAP) questionnaire is an 18-item self-report inventory that was created to disentangle state-wise motivational and consummatory components of everyday activities over a 24-hour period. This scale was used to assess self-reported changes in symptoms of anhedonia before and after inflammation blockade. Respondents respond to statements about daily activities on a scale from 0 (no pleasure/not at all) to 4 (extreme pleasure/very often). Total scores range from 0 to 72 where higher scores indicate greater motivation and effort given to everyday situations.
Time Frame: as for outcome 9
Population: This analysis includes participants who completed this assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sinemet/Placebo | Placebo/Sinemet
Number analyzed (Participants) | 10 | 7
score on a scale
  Visit 1: Pre drug/placebo | 25.5 (11.5) | 26.6 (13.8)
  Visit 1: 1-2 hrs post drug/placebo | 26.9 (11.1) | 25.4 (16.1)
  Visit 2: Pre drug/placebo | 28.9 (13.6) | 25.1 (22.0)
  Visit 2: 1-2 hrs post drug/placebo | 29.2 (13.7) | 25.1 (21.3)

15. Other Pre Specified Outcome: Correlation Coefficient Between Change in Cerebral Blood Flow (CBF) and Change in Functional Connectivity
Description: The cerebral blood flow (CBF) before and after Sinemet (250 mg levodopa/ 50mg carbidopa) or placebo administration was assessed by arterial spin labeling (ASL) fMRI.
Time Frame: Scans approximately 45 minutes post drug/placebo administration at Visit 1, Visit 2 (spaced by approximately 1 week)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From time of consent until follow up (up to 2 weeks).
Description: The population analyzed includes all subjects who were randomized and had taken at least one dose of the medication.
Groups:
- Sinemet: Levodopa+carbidopa (Sinemet) is a combination of 250 mg levodopa and 50 mg carbidopa. Sinemet was administered orally either at Visit 1 if the subject was in the Sinemet/Placebo group or, at Visit 2 if the subject was in the Placebo/Sinemet group.
- Placebo: Placebo: A placebo is a sugar pill that has no therapeutic effect and was administered orally either at Visit 1 if the subject was in the Placebo/Sinemet group or, at Visit 2 if the subject was in the Sinemet/Placebo group.
Arm/Group | Sinemet | Placebo
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 50/57 | 11/56
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sinemet (N=57) | Placebo (N=56)
Headache (Nervous system disorders) | 6 (6) | 5 (5)
Vomiting (Gastrointestinal disorders) | 8 (9) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 22 (27) | 3 (3)
Lightheadedness (General disorders) | 5 (5) | 0 (0)
Feeling Hot (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02513485/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT02513485/ICF_001.pdf